CLINICAL TRIAL: NCT05924789
Title: Epidemiological Characteristics of Gastric and Pancreatic Cancers in Latin America
Acronym: GASPAR
Status: Completed | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Astellas Pharma Inc (Industry); Grupo Argentino de Investigación Clínica en Oncología (GAICO) (Unknown)
Responsible Party: Sponsor
Other Study IDs: LACOG0222
Record Dates: First submitted 2023-03-08; First posted 2023-06-29 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Gastric Cancer; GastroEsophageal Cancer; Pancreatic Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: 120 patients with histological diagnosis of gastric and gastroesophageal junction cancer.
  Interventions: Other: Observational study
- Cohort B: 80 patients histological diagnosis of pancreatic cancer.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — This is an observational study; patients will not be exposed to clinical interventions different from those belonging to the standard of care.

SUMMARY:
Currently, there is no Brazilian or Latin American epidemiological data, such as clinical-pathological characteristics, standard treatments and outcomes of gastric cancer and pancreatic cancer in the region. The study aims to create a Latin American multicenter database to analyze epidemiological, clinical, and pathological data, treatments, outcomes, and biological information from patients with gastric and pancreatic cancer.

DETAILED DESCRIPTION:
Patients diagnosed with gastric and gastroesophageal junction or pancreatic cancer after January 2019 at participating sites will be included. Data will be collected from medical records in selected centers that comprise different countries from Latin America. Data collection will begin on the time of site activation.

Patients recruited for this study will be identified in the participating sites. Data from clinical, demographic, and socioeconomic variables will be collected. Also, data on treatments performed and outcomes will be abstracted. The patient data sources will be the medical records of the patients. Patients will continue to receive treatment and clinical evaluations for gastric and gastroesophageal junction or pancreatic cancer according to what is determined by their medical team, according to the usual standards of treatment and clinical practice of each center.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* Histological diagnosis of gastric and gastroesophageal junction cancer (Cohort A) or histological diagnosis of pancreatic cancer (Cohort B);
* Advanced disease diagnosis from January 2019: patients can be included prospectively. Advanced disease is defined as metastatic disease or locally advanced disease not amenable to curative therapy;
* Availability of adequate medical data for data collection.

Exclusion Criteria:

* Synchronous invasive tumor or second primary tumor in the last three years (except thyroid tumors or non-melanoma skin);
* Nonepithelial histology in Cohort A: Sarcoma, GIST, lymphoma, and tumors of neuroendocrine origin;
* Nonepithelial histology in Cohort B: Sarcoma, GIST, lymphoma, pancreatoblastoma, and tumors of neuroendocrine origin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastric and gastroesophageal junction or pancreatic cancer after January 2019.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-08-11 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Describe the treatment patterns | During study duration (one year)
  Describe the treatment patterns and outcomes of patients with gastric and gastroesophageal junction cancer in Latin America.

CONTACTS AND LOCATIONS:
Overall Officials: Renata D´Alpino Peixoto, Principal Investigator — Latin American Cooperative Oncology Group
Locations (6):
- Instituto de Oncología San Gerónimo, Santa Fe, Santa Fe Province, Argentina
- Brazil (5):
  - ÉTICA Clínica AMO - Assistência Multidisciplinar em Oncologia, Salvador, Estado de Bahia
  - HMV - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CEPON - Centro de Pesquisas Oncológicas, Florianópolis, Santa Catarina
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - A.C. Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: No